CLINICAL TRIAL: NCT00231257
Title: A Multicenter, Randomized Study of the Sirolimus-Eluting Bx VELOCITY® BALLOON Expandable Stent vs. Intravascular Brachytherapy in the Treatment of Patients With In-Stent Restenotic Coronary Artery Lesions
Brief Title: Sirolimus-Eluting Stent vs. Intravascular Brachytherapy in In-Stent Restenotic Coronary Artery Lesions(SISR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: David R. Holmes, Jr., MD, Mayo Clinic Rochester, Minnesota
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P02-6313
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: In-Stent Restenosis
MeSH Terms: interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cypher Bx Velocity
  Interventions: Device: Sirolimus-Eluting Bx Velocity® Balloon Expandable Stent
- 2 (Active Comparator): Brachytherapy
  Interventions: Procedure: Brachytherapy

INTERVENTIONS:
Device: Sirolimus-Eluting Bx Velocity® Balloon Expandable Stent — Sirolimus-Eluting Bx Velocity® Balloon Expandable Stent
  Arms: 1
Procedure: Brachytherapy — Brachytherapy
  Arms: 2

SUMMARY:
The main objective of this study is to demonstrate the superiority or non-inferiority of the sirolimus-eluting Bx VELOCITY® stent compared to intravascular brachytherapy in patients with in-stent restenotic native coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient has an in-stent restenosis of > 50% (by subjective angiographic determination of the minimal luminal diameter compared to the distal reference diameter) within a native coronary artery which has previously undergone stent placement ( 4 weeks). Lesions must meet ISR Classification I-III.

  2. The patient has a history, signs of, or laboratory studies that suggest coronary ischemia attributable to the target stenosis. The diagnosis of angina pectoris is defined by Canadian Cardiovascular Society Classification (CCS I, II, III, or IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II) OR patients with documented silent ischemia;

  3. The study target lesion must be located in an in-stent restenotic native coronary artery measuring > 2.75mm and 3.5mm in diameter and > 15mm and 40mm in length to allow treatment with a maximum of three 18mm stents. The target lesion must have undergone coronary interventional treatment > 4 weeks previously. Patients with one or more prior percutaneous coronary interventions at the target lesion are acceptable candidates.

  4. The vessel 1cm distal to the target lesion is > 2.5mm in diameter;

  5. Ejection Fraction must be > 40%;

  6. The study target lesion cannot be located in a vessel containing a second lesion requiring treatment at the time of the procedure.

  7. Male or non-pregnant female patients > 18 years of age inclusive. NOTE: Females of child-bearing potential must have a negative pregnancy test (urine or serum) prior to enrollment and must use birth control for 6 months.

Exclusion Criteria:

1. The study target lesion has definite or possible thrombus present by angiographic criteria.
2. The patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK > 2 times normal within the preceding 24 hours and the CK and CK-MB enzymes remain above normal at the time of treatment.
3. Impaired renal function (Serum creatinine > 2.0mg/dl);
4. The patient has unstable angina classified as Braunwald III B or C, or is having peri infarction angina.
5. The left ventricular ejection fraction is < 40%.
6. The target vessel has previously sustained a perforation.
7. Totally occluded vessel (TIMI 0 level);
8. Prior stent within 5mm of target lesion;
9. There is a total occlusion of the restenosed-stent (ISR Classification IV) prior to the interventional procedure.
10. Has an ostial target lesion;
11. Significant (> 50%) in-stent restenoses proximal or distal to the target lesion that might require revascularization or impede runoff;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2003-02; Primary Completion 2005-01 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Target vessel failure (TVF) defined as cardiac death, myocardial infarction, or target vessel revascularization at 9 months post-procedure. | 9 months post-procedure.

SECONDARY OUTCOMES:
Angiographic in-lesion and in-stent binary restenosis (³ 50% diameter stenosis) at 6 months post-procedure (by QCA). | 6 months post-procedure
Post-procedure and six-month in-stent and in-lesion percent diameter stenosis (%DS) and late loss at 6 months post-procedure (by QCA) - [analysis at 6 months chosen so that results from the GAMMA Trial can be used]. | 6 months post-procedure
Post-procedure and six-month in-stent and in-lesion minimum lumen diameter (MLD) (by QCA). | Post-procedure and at six-month
Target lesion revascularization (TLR) at 6 and 9 months post-procedure. | 6 and 9 months post-procedure
Target vessel revascularization (TVR) at 6 and 9 months post-procedure. | 6 and 9 months post-procedure
Composite of Major Adverse Cardiac Events (MACE) defined as death, myocardial infarction (Q wave and non-Q wave), emergent bypass surgery, or repeat target lesion revascularization at 30 days and 6, 9, and 12-months, and 2, 3, 4, and 5 years post-proce | 30 days and 6, 9, and 12-months, and 2, 3, 4, and 5 years post-procedure
Stent lumen and stent obstruction volume by intravascular ultrasound (IVUS) at post-procedure and six months in a subset of patients conducted at 5-7 investigational centers. | post-procedure and six months
Cost associated with the index hospitalization, length of stay, and repeat hospitalizations during the 12 mo post-procedure follow-up. | 12 mo post-procedure
Rate of late thrombosis | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: David R. Holmes, Jr., MD, Principal Investigator — Mayo Clinic - Rochester, Minnesota
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Holmes DR Jr, Teirstein P, Satler L, Sketch M, O'Malley J, Popma JJ, Kuntz RE, Fitzgerald PJ, Wang H, Caramanica E, Cohen SA; SISR Investigators. Sirolimus-eluting stents vs vascular brachytherapy for in-stent restenosis within bare-metal stents: the SISR randomized trial. JAMA. 2006 Mar 15;295(11):1264-73. doi: 10.1001/jama.295.11.1264. Epub 2006 Mar 12. PMID 16531619
- [Result] Holmes DR Jr, Teirstein PS, Satler L, Sketch MH Jr, Popma JJ, Mauri L, Wang HP, Schleckser PA, Cohen SA; SISR Investigators. 3-year follow-up of the SISR (Sirolimus-Eluting Stents Versus Vascular Brachytherapy for In-Stent Restenosis) trial. JACC Cardiovasc Interv. 2008 Aug;1(4):439-48. doi: 10.1016/j.jcin.2008.05.010. PMID 19463342